CLINICAL TRIAL: NCT02515799
Title: A Double-blind, Placebo Controlled, Randomized Crossover Trial to Characterize the Mucolytic Effectiveness of Tacholiquine® in Chronic Bronchitis
Brief Title: Mucolytic Effectiveness of Tacholiquine ® in Chronic Bronchitis
Acronym: Tacho-COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: bene-Arzneimittel GmbH (Industry)
Collaborators: Medaimun GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 268/14
Record Dates: First submitted 2015-07-24; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive | interventions — tacholiquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacholiquine (Active Comparator): Inhalation
  Interventions: Drug: Tacholiquine
- Saline Solution 0,9% (Placebo Comparator): Inhalation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tacholiquine — Inhaled Tacholiquine ®1% - 5ml
  Arms: Tacholiquine
Other: Placebo — Inhaled Placebo
  Other Names: isotonic saline solution (0.9%)
  Arms: Saline Solution 0,9%

SUMMARY:
The purpose of this study is to evaluate the mucolytic activity of Tacholiquine® compared to saline (0.9%) in chronic bronchitis patients. Lung function parameters, biomarker profiles in sputum and serum, and clinical symptoms by standardized questionnaires [COPD activity index (CAT), Baseline Dyspnea Index (BDI) & Transition Dyspnea Index (TDI)and the St. George's Respiratory Questionnaire (SGRQ)] will be evaluated in response to Tacholiquine® vs. saline in chronic bronchitis patients.

DETAILED DESCRIPTION:
The aim of the study is to compare Tacholiquine ® and saline (0.9%) regarding their ability to promote the discharge of mucus from the respiratory passages in patients with chronic bronchitis (COPD). Alleviated discharge of mucus should ease breathing, improve subjective wellbeing, reduce inflammation in the air passages and improve lung function.

Determine the magnitude of the effect of Tacholiquine ® compared to saline (0.9%) in chronic bronchitis patients. Lung function parameters, biomarker profiles in sputum and serum, and clinical symptoms and quality of life by standardized questionnaires [COPD activity index (CAT), Baseline Dyspnea Index (BDI) & Transition Dyspnea Index (TDI), St George's respiratory Quality of Life Questionnaire] will be evaluated in response to Tacholiquine ® vs. saline at day one and at end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Female or male subjects aged 40-85 years inclusive at Visit 1.
3. Documented history of COPD with a post-bronchodilator FEV1/FVC<0.70 and a post-bronchodilator FEV1<80% of predicted normal value at screening (spirometry will be used for this criteria assessment).
4. Current smoker or ex-smoker with a tobacco history of ≥10 pack-years (1 pack year = 20 cigarettes smoked per day for 1 year).
5. Women of childbearing potential (WOCBP) must use a highly effective form of birth control (confirmed by the Investigator).

   - Women >50 years old would be considered postmenopausal
6. At least a CAT value > 10 at Visit 1.
7. Presence of chronic cough and sputum production either "several days per week" or "almost every day"

Exclusion Criteria:

1. Clinically important pulmonary disease other than COPD (e.g. active lung infection, clinically significant bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency and primary ciliary dyskinesia) or another diagnosed pulmonary or systemic disease that is associated with elevated peripheral eosinophil counts (e.g. allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome).
2. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   * Affect the safety of the subject throughout the study
   * Influence the findings of the study or their interpretation
   * Impede the subject's ability to complete the entire duration of study
3. Documented Unstable ischemic heart disease, arrhythmia, cardiomyopathy, heart failure, renal failure, uncontrolled hypertension as defined by the Investigator, or any other relevant cardiovascular disorder as judged by the Investigator that in Investigator's judgment may put the patient at risk or negatively affect the outcome of the study.
4. Treatment with systemic corticosteroids and/or antibiotics, and/or hospitalization for a COPD exacerbation within 4 weeks prior to (Visit 1).
5. Acute upper or lower respiratory infection requiring antibiotics or antiviral medication within 4 weeks prior to (Visit 1).
6. Pneumonia within 4 weeks prior to (Visit 1), based on the last day of antibiotic treatment or hospitalization date, whatever occurred later. The subject cannot be re-screened if this exclusion criterion is met.
7. History of anaphylaxis to Tacholiquine®.
8. Long term oxygen therapy (LTOT) defined as need for oxygen > 4L 02 flow with signs and/or symptoms of cor pulmonale, right ventricular failure or evidence by echocardiogram or pulmonary artery catheterization of moderate to severe pulmonary hypertension. In order to be admitted to the trial subjects on LTOT have to be ambulatory and be able to attend clinic visits.
9. Any clinically significant abnormal findings in physical examination, vital signs, hematology, or urinalysis during Visit 1, which, in the opinion of the Investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to complete entire duration of the study.
10. Use of immunosuppressive medication, including rectal corticosteroids, high potency topical corticosteroids and systemic steroids within 28 days prior to (Visit 1).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change of sputum weight before, during and after treatment | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  Active Treatment for 3 weeks compared with Placebo (Saline solution 0.9%), 3 inhalations with 5 ml solution via nebulizer per day of study treatment during 21 consecutive days

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  Symptom Score
Baseline Dyspnoea Index (BDI) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  Symptom Score
transition dyspnoea index (TDI) | Visit 1 (day 0), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 6 (day 21±3 after Visit 4)
  Symptom Score
ease of sputum production | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  Ease is measured by analog scale
Change in Forced vital capacity (FVC) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  lung function parameter
change in forced expiratory volume at one second (FEV1) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  lung function parameter
Forced Expiratory Flow at 75% (FEF25) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  lung function parameter
Residual Volume (RV) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  lung function parameter
Ratio of Residual Volume to Total Lung Capacity( RV/TLC) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  lung function parameter
Sputum biomarker profiles (IL-1, IL-6, IL-8) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
CrP | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  Plasma biomarker profile
Lipopolysaccharide-binding protein (LBP) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  Plasma biomarker profile
Interleukin 6 (IL-6) | Visit 1 (day 0), Visit 2 (day 7 ±1), Visit 3 (day 21±3), Visit 4 (day 28±3), Visit 5 (day 7±1 after Visit 4), Visit 6 (day 21±3 after Visit 4)
  Plasma biomarker profile

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof MD, Principal Investigator — Medaimun GmbH
Locations (1):
- Medaimun GmbH, Frankfurt/M, Hesse, Germany

REFERENCES:
- [Background] Decramer M, Janssens W. Mucoactive therapy in COPD. Eur Respir Rev. 2010 Jun;19(116):134-40. doi: 10.1183/09059180.00003610. PMID 20956182
- [Result] Paez PN, Miller WF. Surface active agents in sputum evacuation: a blind comparison with normal saline solution and distilled water. Chest. 1971 Oct;60(4):312-7. doi: 10.1378/chest.60.4.312. No abstract available. PMID 4940230
- [Result] Eickmeier O, Huebner M, Herrmann E, Zissler U, Rosewich M, Baer PC, Buhl R, Schmitt-Grohe S, Zielen S, Schubert R. Sputum biomarker profiles in cystic fibrosis (CF) and chronic obstructive pulmonary disease (COPD) and association between pulmonary function. Cytokine. 2010 May;50(2):152-7. doi: 10.1016/j.cyto.2010.02.004. Epub 2010 Feb 23. PMID 20181491
- [Derived] Koppitz M, Eschenburg C, Salzmann E, Rosewich M, Schubert R, Zielen S. Mucolytic Effectiveness of Tyloxapol in Chronic Obstructive Pulmonary Disease - A Double-Blind, Randomized Controlled Trial. PLoS One. 2016 Jun 16;11(6):e0156999. doi: 10.1371/journal.pone.0156999. eCollection 2016. PMID 27308826